CLINICAL TRIAL: NCT02607800
Title: A Phase 3, Global, Multicenter, Randomized, Open-Label Study to Investigate the Safety and Efficacy of Sofosbuvir/Velpatasvir/GS-9857 Fixed-Dose Combination for 8 Weeks Compared to Sofosbuvir/Velpatasvir for 12 Weeks in Direct-Acting Antiviral-Naïve Subjects With Chronic HCV Infection
Brief Title: Safety and Efficacy of Sofosbuvir/Velpatasvir/Voxilaprevir and Sofosbuvir/Velpatasvir in Adults With Chronic HCV Infection Who Have Not Previously Received Treatment With Direct-Acting Antiviral Therapy
Acronym: POLARIS-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-367-1172; 2015-003460-36 (EudraCT Number)
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C
Keywords: Chronic Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir velpatasvir voxilaprevir drug combination; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SOF/VEL/VOX (Experimental): SOF/VEL/VOX tablet for 8 weeks
  Interventions: Drug: SOF/VEL/VOX
- SOF/VEL 12 weeks (Active Comparator): SOF/VEL tablet for 12 weeks
  Interventions: Drug: SOF/VEL

INTERVENTIONS:
Drug: SOF/VEL/VOX — 400/100/100 mg tablet administered orally once daily with food
  Other Names: GS-7977/GS-5816/GS-9857; Vosevi®
  Arms: SOF/VEL/VOX
Drug: SOF/VEL — 400/100 mg tablet administered orally once daily with or without food
  Other Names: GS-7977/GS-5816; Epclusa®
  Arms: SOF/VEL 12 weeks

SUMMARY:
The primary objectives of this study are to compare the efficacy, safety, and tolerability of treatment with sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX) fixed dose combination (FDC) for 8 weeks with that of SOF/VEL FDC for 12 weeks in direct-acting antiviral-naive participants with chronic hepatitis C virus (HCV) infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent
* HCV RNA ≥ 10^4 IU/mL at screening
* Chronic HCV infection (≥ 6 months)
* HCV treatment naive or treatment experienced with an interferon (IFN)-based regimen
* Use of protocol specified methods of contraception

Key Exclusion Criteria:

* Current or prior history of clinically significant illness that may interfere with participation in the study
* Screening ECG with clinically significant abnormalities
* Laboratory parameters outside the acceptable range at screening
* Pregnant or nursing female
* Chronic liver disease not caused by HCV
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 943 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2016-10-10 (Actual); Study Completion 2017-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (93):
- United States (47):
  - Long Beach, California
  - Los Angeles, California
  - Palo Alto, California
  - Pasadena, California
  - Rialto, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Bastrop, Louisiana
  - Baltimore, Maryland
  - Catonsville, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Hillsborough, New Jersey
  - Manhasset, New York
  - New York, New York
  - The Bronx, New York
  - Asheville, North Carolina
  - Fayetteville, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Houston, Texas
  - Live Oak, Texas
  - San Antonio, Texas
  - Murray, Utah
  - Falls Church, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Australia (5):
  - Darlinghurst, New South Wales
  - Herston, Queensland
  - Fitzroy, Victoria
  - Melbourne, Victoria
  - Perth, Western Australia
- Canada (7):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Brampton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (20):
  - Bobigny
  - Clermont-Ferrand
  - Clichy
  - Créteil
  - Grenoble
  - Lille
  - Limoges
  - Lyon
  - Marseille
  - Montpellier
  - Nice
  - Orléans
  - Paris
  - Pessac
  - Rennes
  - Rouen
  - Strasbourg
  - Toulouse
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (6):
  - Berlin
  - Bonn
  - Cologne
  - Frankfurt am Main
  - Hamburg
  - Hanover
- New Zealand (2):
  - Christchurch
  - Grafton
- San Juan, Puerto Rico
- United Kingdom (5):
  - London
  - Manchester
  - Nottingham
  - Oxford
  - Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/about/ethics-and-code-of-conduct/policies.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/about/ethics-and-code-of-conduct/policies

REFERENCES:
- [Result] Jacobson IM, Asselah T, Nahass R, Bhandari BR, Tran A, Hyland RH, et al. A Randomized Phase 3 Trial of Sofosbuvir/Velpatasvir/Voxilaprevir for 8 Weeks Compared to Sofosbuvir/Velpatasvir for 12 Weeks in DAA-Naïve Genotype 1-6 HCV-Infected Patients: The POLARIS-2 Study [Abstract LB-12]. Hepatology AASLD Abstracts 2016;64 (6 (suppl)):1126A.
- [Result] Jacobson IM, Lawitz E, Gane EJ, Willems BE, Ruane PJ, Nahass RG, Borgia SM, Shafran SD, Workowski KA, Pearlman B, Hyland RH, Stamm LM, Svarovskaia E, Dvory-Sobol H, Zhu Y, Subramanian GM, Brainard DM, McHutchison JG, Brau N, Berg T, Agarwal K, Bhandari BR, Davis M, Feld JJ, Dore GJ, Stedman CAM, Thompson AJ, Asselah T, Roberts SK, Foster GR. Efficacy of 8 Weeks of Sofosbuvir, Velpatasvir, and Voxilaprevir in Patients With Chronic HCV Infection: 2 Phase 3 Randomized Trials. Gastroenterology. 2017 Jul;153(1):113-122. doi: 10.1053/j.gastro.2017.03.047. Epub 2017 Apr 5. PMID 28390869

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Europe, and, Asia Pacific. The first participant was screened on 16 November 2015. The last study visit occurred on 11 January 2017.
Pre-assignment Details: 1116 participants were screened.
Groups:
- SOF/VEL/VOX 8 Weeks: Sofosbuvir/Velpatasvir/Voxilaprevir (Vosevi®; SOF/VEL/VOX) (400/100/100 mg) fixed dose combination (FDC) tablet orally once daily with food for 8 weeks
- SOF/VEL 12 Weeks: Sofosbuvir/Velpatasvir (Epclusa®; SOF/VEL) (400/100 mg) FDC tablet orally once daily with or without food for 12 weeks
Period: Overall Study
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Started | 502 | 441
Completed | 492 | 430
Not Completed | 10 | 11
Not completed — Lost to Follow-up | 7 | 10
Not completed — Withdrew Consent | 2 | 0
Not completed — Randomized/Enrolled but Not Treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who took at least 1 dose of the study drug
Groups:
- SOF/VEL/VOX 8 Weeks: SOF/VEL/VOX (400/100/100 mg) FDC tablet orally once daily with food for 8 weeks
- SOF/VEL 12 Weeks: SOF/VEL (400/100 mg) FDC tablet orally once daily with or without food for 12 weeks
- Total: Total of all reporting groups
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks | Total
Number analyzed (Participants) | 501 | 440 | 941
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (11.1) | 52 (11.9) | 52 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246 | 203 | 449
  Male | 255 | 237 | 492
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 391 | 365 | 756
  Black or African American | 48 | 47 | 95
  Asian | 51 | 22 | 73
  Other | 5 | 2 | 7
  American Indian or Alaska Native | 3 | 2 | 5
  Native Hawaiian or Pacific Islander | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 52 | 84
  Not Hispanic or Latino | 469 | 388 | 857
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 13 | 13 | 26
  Canada | 36 | 24 | 60
  United States | 283 | 269 | 552
  United Kingdom | 24 | 23 | 47
  Australia | 13 | 11 | 24
  France | 105 | 82 | 187
  Germany | 27 | 18 | 45
IL28b Status [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 166 | 136 | 302
    CT | 253 | 245 | 498
    TT | 82 | 59 | 141
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.1 (0.75) | 6.2 (0.66) | 6.2 (0.71)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 155 | 138 | 293
  ≥ 800,000 IU/mL | 346 | 302 | 648

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: all randomized/enrolled participants who took at least 1 dose of the study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 501 | 440
percentage of participants | 95.2 [93.0 to 96.9] | 98.2 [96.4 to 99.2]
Statistical Analysis 1: Comparison: SOF/VEL/VOX 8 Weeks vs SOF/VEL 12 Weeks; Test type: Non-Inferiority — Noninferiority was demonstrated if the lower bound of the 2-sided 95% confidence interval (CI) for the difference in SVR12 was greater than -5%. If the lower bound of the CI was greater than -5% (ie, the noninferiority null hypothesis was rejected), a 2-sided stratified Cochran-Mantel-Haenszel test was to be used to test for the superiority of SOF/VEL/VOX for 8 weeks over SOF/VEL for 12 weeks at a significance level of 0.05; Difference in proportions = -3.2, 95% CI 2-sided [-6.0 to -0.4] — Difference in proportions between treatment groups and associated 95% CI were calculated based on stratum-adjusted Mantel-Haenszel proportions

2. Primary Outcome: Percentage of Participants Who Permanently Discontinue Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 501 | 440
percentage of participants | 0 | 0.5

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOF/VEL/VOX 8 Weeks: SOF/VEL/VOX (400/100/100 mg) tablet orally once daily with food for 8 weeks
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 501 | 440
percentage of participants
  SVR4 | 96.4 [94.4 to 97.9] | 98.9 [97.4 to 99.6]
  SVR 24 | 95.0 [92.7 to 96.7] | 98.0 [96.2 to 99.1]

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ On Treatment
Time Frame: Weeks 1, 2, 4, 8, and 12
Population: Percentage of participants in Full Analysis Set with on-treatment data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 501 | 440
percentage of participants
  Week 1 | 24.8 [21.0 to 28.8] | 22.7 [18.9 to 26.9]
  Week 2: number analyzed (Participants) | 501 | 439
  Week 2 | 65.9 [61.5 to 70.0] | 61.3 [56.5 to 65.9]
  Week 4: number analyzed (Participants) | 501 | 439
  Week 4 | 92.4 [89.7 to 94.6] | 92.0 [89.1 to 94.4]
  Week 8: number analyzed (Participants) | 500 | 439
  Week 8 | 99.2 [98.0 to 99.8] | 99.8 [98.7 to 100.0]
  Week 12: number analyzed (Participants) | 0 | 439
  Week 12 |  | 99.8 [98.7 to 100.0]

5. Secondary Outcome: Change From Baseline in HCV RNA
Time Frame: Baseline; Weeks 1, 2, 4, 8, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 501 | 440
log10 IU/mL
  Week 1: number analyzed (Participants) | 491 | 433
  Week 1 | -4.23 (0.689) | -4.24 (0.679)
  Week 2: number analyzed (Participants) | 496 | 436
  Week 2 | -4.75 (0.747) | -4.77 (0.646)
  Week 4: number analyzed (Participants) | 501 | 437
  Week 4 | -4.95 (0.750) | -4.99 (0.656)
  Week 8: number analyzed (Participants) | 496 | 439
  Week 8 | -4.99 (0.754) | -5.03 (0.655)
  Week 12: number analyzed (Participants) | 0 | 438
  Week 12 |  | -5.03 (0.656)

6. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
Number analyzed (Participants) | 501 | 440
percentage of participants | 4.2 | 0.7

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF/VEL/VOX 8 Weeks | SOF/VEL 12 Weeks
All-Cause Mortality (participants affected / at risk) | 0/501 | 0/440
Serious Adverse Events (participants affected / at risk) | 15/501 | 7/440
Other Adverse Events (participants affected / at risk) | 280/501 | 213/440
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX 8 Weeks (N=501) | SOF/VEL 12 Weeks (N=440)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Perineal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL/VOX 8 Weeks (N=501) | SOF/VEL 12 Weeks (N=440)
Diarrhoea (Gastrointestinal disorders) | 88 | 32
Nausea (Gastrointestinal disorders) | 80 | 40
Asthenia (General disorders) | 32 | 27
Fatigue (General disorders) | 106 | 91
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 24
Headache (Nervous system disorders) | 134 | 99
Insomnia (Psychiatric disorders) | 26 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years